CLINICAL TRIAL: NCT01262274
Title: Randomized Phase II Trial of Anastrozole in Combination With/Without Metronomic Tegafur-uracil as Neo-adjuvant Therapy in Postmenopausal Primary Breast Cancer
Brief Title: Randomized Phase II Trial of Anastrozole Plus Metronomic Tegafur-uracil as Neo-adjuvant Therapy in Postmenopausal Breast Cancer
Acronym: Neo-ACET BC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to an adverse event revelation.
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Department of breast and endocrine surgery graduate school of Medicine Osaka University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIBC1009
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ANA (Active Comparator)
  Interventions: Drug: Anastrozole
- ANA+UFT (Experimental)
  Interventions: Drug: Anastrozole plus tegafur-uracil

INTERVENTIONS:
Drug: Anastrozole — ANA is given 1mg daily for 24 weeks.
  Arms: ANA
Drug: Anastrozole plus tegafur-uracil — ANA is given 1mg daily for 24 weeks. UFT is given by 270mg/m2 twice a day for 24 weeks.
  Arms: ANA+UFT

SUMMARY:
The Aim of this study is to validate a treatment of anastrozole in combination with tegafur-uracil as pre-operative therapy for postmenopausal primary breast cancer. Although pre-operative hormone therapy is a novel therapeutic approach, only hormone therapy has limitation in terms of efficacy. Metronomic chemotherapy, which is the frequent administration of low-dose cytotoxic agents, is not only target tumor cells but also inhibiting angiogenesis. Because there was a report that efficacy of hormone therapy add to metronomic chemotherapy as pre-operative therapy, a randomized phase II trial of anastrozole (ANA) in combination with/without metronomic tegafur-uracil (UFT) as neo-adjuvant for postmenopausal breast cancer will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of invasive breast cancer
* Clinical stage T2, N0 or N1, M0 (TNM Classification)
* Patients must be postmenopausal
* Tumors are estrogen receptor (ER) positive and human epidermal growth factor receptor (HER2) negative
* ECOG Performance status (PS) 0 or 1
* Patients must be able to swallow tablets and capsules
* Candidates for mastectomy or breast-conserving surgery
* Adequate bone marrow, liver and renal function
* Written informed consent was obtained from all patients before randomization.

Exclusion Criteria:

* Inoperable, bilateral or inflammatory breast cancer
* multiple carcinoma
* Personal history of invasive carcinoma
* Patients receive systemic therapy of corticosteroid
* Patients receive estrogen preparation or raloxifene
* Patients with other concurrent severe and/or uncontrolled medical disease
* Patients whom doctors judged inadequate to the enrollment of this study by other reasons.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Response Rate (confirmed by calipers CT or MRI) | six months

SECONDARY OUTCOMES:
Reduction Rate, Pathological response, Breast-conserving surgery rate, Adverse event rate, Predictive factor | seven months

CONTACTS AND LOCATIONS:
Overall Officials: Shinzaburo Noguchi, M.D., Ph.D., Principal Investigator — Department of Breast and Endocrine Surgery, Osaka University Graduate School of Medicine
Locations (1):
- Department of Breast and Endocrine Surgery, Osaka University Graduate School of Medicine, Osaka, Osaka, Japan